CLINICAL TRIAL: NCT04306718
Title: Cultivation of Hyalocytes From ILM and ERM Samples: a Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of department, Professor, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: hya
Record Dates: First submitted 2019-10-21; First posted 2020-03-13 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- studyarm (Experimental): Hyalocytes from ERM and ILM are cultured in alphaMEM to examine their proliferation habits
  Interventions: Procedure: membrane peeling

INTERVENTIONS:
Procedure: membrane peeling — ERM and ILM are peeled routinely during surgery

SUMMARY:
ILM and ERM are routinely excised during surgery, as part of the surgical technique, and cultivation of hyalocytes will be performed ex vivo after surgery.

DETAILED DESCRIPTION:
Hyalocytes, typically located 20 to 50μm anterior the internal limiting membrane (ILM), have the potential to contribute to development of epiretinal membranes (ERM) in presence of vitreoschisis. For macular holes, hyalocytes located on the ILM are hypothesized to contribute to the closure of the macular hole after application of the inverted ILM flap technique.

ILM is routinely excised during surgical repair of macular holes. During peeling of ERM it is excised in case of persisting wrinkling of the retinal surface or partial en bloc excision with the ERM. Furthermore, excision of ILM during ERM peeling is associated with significantly lower recurrence rates of ERM and better Long term visual acuity, according to the results reported by Chang et al. Removal of ERM and ILM is part of the surgical routine during surgical repair of macular holes and peeling of epiretinal membranes. Therefore, cultivation of excised ERM and ILM samples does not increase risks for patients in any way. During study it is planned to cultivate hyalocytes for investigation of their role in macular hole closure.

ELIGIBILITY:
Inclusion Criteria:

* Macular hole or epiretinal Membrane

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proliferation of Hyalocytes | 9 days
  hyalocytes from ERM and ILM will be cultured and counted

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Dr., Principal Investigator — VIROS at Hanuschkrankenhaus
Locations (1):
- VIROS at Hanuschkrankenhaus, Vienna, Austria

REFERENCES:
- [Background] Chang WC, Lin C, Lee CH, Sung TL, Tung TH, Liu JH. Vitrectomy with or without internal limiting membrane peeling for idiopathic epiretinal membrane: A meta-analysis. PLoS One. 2017 Jun 16;12(6):e0179105. doi: 10.1371/journal.pone.0179105. eCollection 2017. PMID 28622372